CLINICAL TRIAL: NCT01746225
Title: A Randomized Phase II Study Evaluating Different Schedules of Nab-Paclitaxel in Metastatic Breast Cancer (SNAP Trial)
Brief Title: Schedules of Nab-Paclitaxel in Metastatic Breast Cancer
Acronym: SNAP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ETOP IBCSG Partners Foundation (Network)
Collaborators: Breast International Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IBCSG 42-12 / BIG 2-12; 2012-003058-10 (EudraCT Number)
Record Dates: First submitted 2012-11-28; First posted 2012-12-10 (Estimated); Results first posted 2020-03-27 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Metastatic Breastcancer
Keywords: Metastatic; Breast; Cancer; HER2-negative Stage IV; No previous chemotherapy
MeSH Terms: conditions — Neoplasm Metastasis; Neoplasms | interventions — 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A: nab-Paclitaxel 150 mg/m2 days 1,15 (Experimental): Arm A: Induction* nab-Paclitaxel 125 mg/m2 on days 1,8,15 every 28 days for 3 cycles followed by maintenance nab-Paclitaxel 150 mg/m2 administered on days 1, 15 of each 28-day cycle (total 300mg/m2 per cycle) until progression or unacceptable toxicity.
  *Following Amendment 1, the dose in the induction phase dose in all three arms was reduced to 125 mg/m² from 150 mg/m².
  Interventions: Drug: nab-Paclitaxel
- B: nab-Paclitaxel 100 mg/m2 days 1,8,15 (Experimental): Arm B: Induction* nab-Paclitaxel 125 mg/m2 on days 1,8,15 every 28 days for 3 cycles followed by maintenance nab-Paclitaxel 100 mg/m2 administered on days 1, 8, 15 of each 28-day cycle (total 300mg/m2 per cycle) until progression or unacceptable toxicity.
  *Following Amendment 1, the dose in the induction phase dose in all three arms was reduced to 125 mg/m² from 150 mg/m².
  Interventions: Drug: nab-Paclitaxel
- C: nab-Paclitaxel 75 mg/m2 days 1,8,15,22 (Experimental): Arm C: Induction* nab-Paclitaxel 125 mg/m2 on days 1,8,15 every 28 days for 3 cycles followed by maintenance nab-Paclitaxel 75 mg/m2 administered on days 1, 8, 15, 22 of each 28-day cycle (total 300mg/m2 per cycle) until progression or unacceptable toxicity.
  *Following Amendment 1, the dose in the induction phase dose in all three arms was reduced to 125 mg/m² from 150 mg/m².
  Interventions: Drug: nab-Paclitaxel

INTERVENTIONS:
Drug: nab-Paclitaxel — Induction phase: 3 cycles of nab-Paclitaxel days 1, 8, 15. Maintenance phase with three maintenance schedules of nab-Paclitaxel (same total dose per cycle, different number of administrations)
  Other Names: Abraxane

SUMMARY:
Longer first line chemotherapy duration has recently been associated with a modest, but significant improvement in overall survival and a clinically meaningful and statistically significant improvement in progression-free survival, in metastatic breast cancer patients. Prolonging chemotherapy until disease progression, however, must be weighed against the detrimental effects of continuous chemotherapy delivery. The SNAP trial seeks to improve the tolerability of prolonged chemotherapy administration strategy by studying alternative treatment schedules, while preserving and possibly improving treatment efficacy in this disease setting.

The availability of a new nanoparticle albumin-bound taxane, nab-Paclitaxel (Abraxane®), represents an opportunity to test this hypothesis. Nab-Paclitaxel has been developed in an attempt to reduce the toxicity associated with standard taxane administration (caused by the use of chemical solvents) while increasing antitumor efficacy.

The SNAP randomized phase II trial evaluates three schedules of nab-Paclitaxel as prolonged chemotherapy administration strategy. Each of three arms will be compared to a historical reference of seven-month median progression-free survival (PFS) based on the most recent trial with docetaxel as control arm to determine whether any of the three arms are worthy of further investigation.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed HER2-negative metastatic (stage IV) breast cancer.
* Measurable or non-measurable, but radiologically evaluable, disease according to RECIST 1.1 criteria.
* Female aged 18 years or older.
* Life expectancy > 3 months.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
* Either ER-positive or ER-negative disease. Patients with ER-positive disease must be endocrine resistant, defined as having failed at least one prior endocrine therapy for breast cancer, or must be candidates for first-line chemotherapy.
* If previously treated with a taxane or anthracycline in the neoadjuvant or adjuvant setting, the period from end of treatment to disease recurrence must have been > 12 months (> 365 days).
* Radiation therapy, if given and regardless of site, must be completed at least 2 weeks prior to randomization.
* Normal hematologic status.
* Normal renal function.
* Normal liver function.
* Normal cardiac function.
* Women of childbearing potential: documented negative pregnancy test within 2 weeks prior to randomization, and acceptable birth control during the duration of the trial therapy and for a period of 6 months following the last administration of study drug.
* Written Informed Consent (IC) must be signed and dated by the patient and the Investigator prior to randomization.
* Completed baseline Quality of Life Form.
* The patient has been informed of and agrees to data transfer and handling, in accordance with national data protection guidelines.
* Availability of an formalin fixed paraffin embedded (FFPE) block from the primary tumor (breast lesion) for submission to central pathology review and for translational research.
* Written consent to pathology material submission, signed and dated by the patient and the Investigator prior to randomization.

Exclusion Criteria:

* Any prior chemotherapy for metastatic breast cancer.
* Presence of central nervous system (CNS) metastasis.
* Peripheral neuropathy grade 2 or higher (CTCAE version 4).
* Significant uncontrolled cardiac disease (i.e. unstable angina, recent myocardial infarction within prior 6 months), patients classified as having a New York Heart Association (NYHA) class III or IV congestive heart failure.
* Pregnant or lactating.
* Prior history of non-breast malignancy (except for adequately controlled basal cell carcinoma of the skin, carcinoma in situ of the cervix, in situ carcinoma of the bladder).
* Any concurrent condition which in the Investigator's opinion makes it inappropriate for the patient to participate in the trial or which would jeopardize compliance with the protocol.
* Contraindications or known hypersensitivity to the study medication or excipients.
* The use of any anti-cancer investigational agents within 30 days prior to expected start of trial treatment.
* Inability or unwillingness to abide by the study protocol or cooperate fully with the Investigator.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2013-04; Primary Completion 2016-05 (Actual); Study Completion 2023-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Gennari, MD, Study Chair — Division of Medical Oncology, E.O. Galliera, Genoa, Italy; Guy Jerusalem, MD, PhD, Study Chair — CHU Sart Tilman and University of Liège, Liège, Belgium
Locations (41):
- Belgium (3):
  - CHR de la Citadelle, Oncology-Haematology Unit, Liège
  - CHU Sart Tilman, Medical Oncology, Liège
  - Centre Hospitalier Peltzer-La Tourelle, Department of Clinical Cancerology, Verviers
- Ireland (10):
  - Bon Secours, Cork
  - Cork University Hospital, Cork
  - Beaumont Hospital, Dublin
  - Mater Misericordiae University Hospital, Dublin
  - Mater Private Hospital, Dublin
  - St James's Hospital, Dublin
  - St Vincent's University Hospital, Dublin
  - University Hospital Galway, Galway
  - Mid-Western Regional Hospital, Limerick
  - Waterford Regional Hospital, Waterford
- Italy (11):
  - Azienda Ospedaliera SS Antonio e Biagio, Alessandria
  - Ospedale degli Infermi, Biella
  - IRCCS MultiMedica, Castellanza
  - E.O. Ospedali Galliera, Genova
  - Istituto Europeo di Oncologia (IEO), Milan
  - Uo Medicina Ocologica Ospedale Di Carpri e Mirandola, Azienda USL di Modena, Modena
  - Fondazione Salvatore Maugeri, Pavia
  - U.O. Oncologia, AUSL Rimini, Rimini
  - Universita degli Studi di Roma La Sapienza, Roma
  - Azienda Osp. Universitaria di Udine, Udine
  - Ospedale di Circolo e Fondatione Macchi, Varese
- Institute of Oncology, Ljubljana, Slovenia
- Spain (5):
  - Hospital Universitari Vall D'Hebron, Barcelona
  - Consorcop Hospitalario Provincial De Castellon, Castelló
  - Hospital Universitari Arnau De Vilanova De Lleida, Lleida
  - Hospital Universitari Sant Joan De Reus, Tarragona
  - Hospital Universitario Lozano Blesa De Zaragoza, Zaragoza
- Switzerland (11):
  - Kantonsspital Aarau, Aarau
  - Universitätsspital Basel, Basel
  - Instituto Oncologico della Svizzera Italiana, Bellinzona
  - Universitätsspital/ Inselspital Bern, Bern
  - Spitalzentrum Biel, Biel
  - Kantonsspital Graubünden, Chur
  - Kantonsspital Baselland, Liestal
  - Luzerner Kantonsspital, Lucerne
  - Kantonsspital St. Gallen, Sankt Gallen
  - Onkologiezentrum Thun-Berner Oberland, Thun
  - Kantonsspital Winterthur, Winterthur

REFERENCES:
- [Background] Chia SK, Speers CH, D'yachkova Y, Kang A, Malfair-Taylor S, Barnett J, Coldman A, Gelmon KA, O'reilly SE, Olivotto IA. The impact of new chemotherapeutic and hormone agents on survival in a population-based cohort of women with metastatic breast cancer. Cancer. 2007 Sep 1;110(5):973-9. doi: 10.1002/cncr.22867. PMID 17647245
- [Background] Gennari A, Conte P, Rosso R, Orlandini C, Bruzzi P. Survival of metastatic breast carcinoma patients over a 20-year period: a retrospective analysis based on individual patient data from six consecutive studies. Cancer. 2005 Oct 15;104(8):1742-50. doi: 10.1002/cncr.21359. PMID 16149088
- [Background] Andre F, Slimane K, Bachelot T, Dunant A, Namer M, Barrelier A, Kabbaj O, Spano JP, Marsiglia H, Rouzier R, Delaloge S, Spielmann M. Breast cancer with synchronous metastases: trends in survival during a 14-year period. J Clin Oncol. 2004 Aug 15;22(16):3302-8. doi: 10.1200/JCO.2004.08.095. PMID 15310773
- [Background] Dawood S, Broglio K, Gonzalez-Angulo AM, Buzdar AU, Hortobagyi GN, Giordano SH. Trends in survival over the past two decades among white and black patients with newly diagnosed stage IV breast cancer. J Clin Oncol. 2008 Oct 20;26(30):4891-8. doi: 10.1200/JCO.2007.14.1168. Epub 2008 Aug 25. PMID 18725649
- [Derived] Gennari A, Sun Z, Hasler-Strub U, Colleoni M, Kennedy MJ, Von Moos R, Cortes J, Vidal MJ, Hennessy B, Walshe J, Parraga KA, Ribi K, Bernhard J, Murillo SM, Pagani O, Barbeaux A, Borstnar S, Rabaglio-Poretti M, Maibach R, Regan MM, Jerusalem G; International Breast Cancer Study Group, Cancer Trials Ireland and SOLTI Group. A randomized phase II study evaluating different maintenance schedules of nab-paclitaxel in the first-line treatment of metastatic breast cancer: final results of the IBCSG 42-12/BIG 2-12 SNAP trial. Ann Oncol. 2018 Mar 1;29(3):661-668. doi: 10.1093/annonc/mdx772. PMID 29228091

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 255 patients were randomized between 16April2013 and 7August2015 at 35 centers in 5 countries.
Groups:
- A: Nab-Paclitaxel 150 mg/m2 Days 1,15: Arm A: Induction* nab-Paclitaxel 125 mg/m2 on days 1,8,15 every 28 days for 3 cycles followed by maintenance nab-Paclitaxel 150 mg/m2 administered on days 1, 15 of each 28-day cycle (total 300mg/m2 per cycle) until progression or unacceptable toxicity.
  nab-Paclitaxel: Induction phase: 3 cycles of nab-Paclitaxel days 1, 8, 15. Maintenance phase with three maintenance schedules of nab-Paclitaxel (same total dose per cycle, different number of administrations)
  *Following Amendment 1, the dose in the induction phase dose in all three arms was reduced to 125 mg/m² from 150 mg/m².
- B: Nab-Paclitaxel 100 mg/m2 Days 1,8,15: Arm B: Induction* nab-Paclitaxel 125 mg/m2 on days 1,8,15 every 28 days for 3 cycles followed by maintenance nab-Paclitaxel 100 mg/m2 administered on days 1, 8, 15 of each 28-day cycle (total 300mg/m2 per cycle) until progression or unacceptable toxicity.
  nab-Paclitaxel: Induction phase: 3 cycles of nab-Paclitaxel days 1, 8, 15. Maintenance phase with three maintenance schedules of nab-Paclitaxel (same total dose per cycle, different number of administrations)
  *Following Amendment 1, the dose in the induction phase dose in all three arms was reduced to 125 mg/m² from 150 mg/m².
- C: Nab-Paclitaxel 75 mg/m2 Days 1,8,15,22: Arm C: Induction* nab-Paclitaxel 125 mg/m2 on days 1,8,15 every 28 days for 3 cycles followed by maintenance nab-Paclitaxel 75 mg/m2 administered on days 1, 8, 15, 22 of each 28-day cycle (total 300mg/m2 per cycle) until progression or unacceptable toxicity.
  nab-Paclitaxel: Induction phase: 3 cycles of nab-Paclitaxel days 1, 8, 15. Maintenance phase with three maintenance schedules of nab-Paclitaxel (same total dose per cycle, different number of administrations)
  *Following Amendment 1, the dose in the induction phase dose in all three arms was reduced to 125 mg/m² from 150 mg/m².
Period: Overall Study
Arm/Group | A: Nab-Paclitaxel 150 mg/m2 Days 1,15 | B: Nab-Paclitaxel 100 mg/m2 Days 1,8,15 | C: Nab-Paclitaxel 75 mg/m2 Days 1,8,15,22
Started | 83 | 86 | 86
Completed | 43 | 40 | 43
Not Completed | 40 | 46 | 43
Not completed — Death | 1 | 0 | 1
Not completed — Withdrawal by Subject | 5 | 15 | 19
Not completed — Physician Decision | 14 | 11 | 3
Not completed — Adverse Event | 15 | 12 | 17
Not completed — Continuing Treatment | 5 | 8 | 3

BASELINE CHARACTERISTICS:
Population: Intention-to-treat population. Arm A had randomized 86 patient, but only 83 were analyzed. 3 patients excluded from analysis, who immediately withdrew consent or cancelled treatment.
Groups:
- A: Nab-Paclitaxel 150 mg/m2 Days 1,15: Arm A: Induction* nab-Paclitaxel 125 mg/m2 on days 1,8,15 every 28 days for 3 cycles followed by maintenance nab-Paclitaxel 150 mg/m2 administered on days 1, 15 of each 28-day cycle (total 300mg/m2 per cycle) until progression or unacceptable toxicity.
  *Following Amendment 1, the dose in the induction phase dose in all three arms was reduced to 125 mg/m² from 150 mg/m².
  nab-Paclitaxel: Induction phase: 3 cycles of nab-Paclitaxel days 1, 8, 15. Maintenance phase with three maintenance schedules of nab-Paclitaxel (same total dose per cycle, different number of administrations)
- B: Nab-Paclitaxel 100 mg/m2 Days 1,8,15: Arm B: Induction* nab-Paclitaxel 125 mg/m2 on days 1,8,15 every 28 days for 3 cycles followed by maintenance nab-Paclitaxel 100 mg/m2 administered on days 1, 8, 15 of each 28-day cycle (total 300mg/m2 per cycle) until progression or unacceptable toxicity.
  *Following Amendment 1, the dose in the induction phase dose in all three arms was reduced to 125 mg/m² from 150 mg/m².
  nab-Paclitaxel: Induction phase: 3 cycles of nab-Paclitaxel days 1, 8, 15. Maintenance phase with three maintenance schedules of nab-Paclitaxel (same total dose per cycle, different number of administrations)
- C: Nab-Paclitaxel 75 mg/m2 Days 1,8,15,22: Arm C: Induction* nab-Paclitaxel 125 mg/m2 on days 1,8,15 every 28 days for 3 cycles followed by maintenance nab-Paclitaxel 75 mg/m2 administered on days 1, 8, 15, 22 of each 28-day cycle (total 300mg/m2 per cycle) until progression or unacceptable toxicity.
  *Following Amendment 1, the dose in the induction phase dose in all three arms was reduced to 125 mg/m² from 150 mg/m².
  nab-Paclitaxel: Induction phase: 3 cycles of nab-Paclitaxel days 1, 8, 15. Maintenance phase with three maintenance schedules of nab-Paclitaxel (same total dose per cycle, different number of administrations)
- Total: Total of all reporting groups
Arm/Group | A: Nab-Paclitaxel 150 mg/m2 Days 1,15 | B: Nab-Paclitaxel 100 mg/m2 Days 1,8,15 | C: Nab-Paclitaxel 75 mg/m2 Days 1,8,15,22 | Total
Number analyzed (Participants) | 83 | 86 | 86 | 255
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 58 [49 to 67] | 56 [45 to 65] | 60 [52 to 68] | 58 [49 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 86 | 86 | 255
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 83 | 85 | 85 | 253
  Asian | 0 | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  Belgium | 10 | 10 | 11 | 33
  Ireland | 21 | 22 | 18 | 61
  Italy | 12 | 16 | 12 | 40
  Slovenia | 3 | 1 | 3 | 7
  Switzerland | 20 | 25 | 29 | 75
  Spain | 17 | 12 | 13 | 42
ER Status [Count of Participants; unit: Participants]
  Positive | 72 | 69 | 69 | 210
  Negative | 11 | 17 | 17 | 45
Prior Taxanes [Count of Participants; unit: Participants]
  Yes | 26 | 28 | 26 | 80
  No | 57 | 58 | 60 | 175
Type of Radiologically Evaluable Disease [Count of Participants; unit: Participants]
  Measurable | 68 | 73 | 69 | 210
  Non-measurable only | 15 | 13 | 17 | 45

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Time from randomization until objective disease progression [progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions] or death, whichever occurs first. For patients without progression, follow-up was censored at the date of last disease assessment without progression, unless death occurred within a short period of time (12 weeks) following the date last known progression-free, in which case the death was counted as a PFS event.
Time Frame: Reported after 18.2 months median follow-up since randomization
Population: Intention-to-treat population
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | A: Nab-Paclitaxel 150 mg/m2 Days 1,15 | B: Nab-Paclitaxel 100 mg/m2 Days 1,8,15 | C: Nab-Paclitaxel 75 mg/m2 Days 1,8,15,22
Number analyzed (Participants) | 83 | 86 | 86
months | 7.9 [6.8 to 8.4] | 9.0 [8.1 to 10.9] | 8.5 [6.7 to 9.5]
Statistical Analysis 1: Comparison: A: Nab-Paclitaxel 150 mg/m2 Days 1,15; For each arm separately, PFS was compared to the historic PFS of first-line docetaxel using a one-sample one-sided log-rank test, of the null hypothesis, H0: median PFS≤7 months vs. H1: median PFS>7 months; Test type: Superiority; p = 0.12, Log Rank — Not adjusted for multiple comparisons; One-sided .05 alpha-level test; One-sided test
Statistical Analysis 2: Comparison: B: Nab-Paclitaxel 100 mg/m2 Days 1,8,15; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .03, Log Rank — Not adjusted for multiple comparisons; One-sided .05 alpha-level test; One-sided test
Statistical Analysis 3: Comparison: C: Nab-Paclitaxel 75 mg/m2 Days 1,8,15,22; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .20, Log Rank — Not adjusted for multiple comparisons; One-sided .05 alpha-level test; One-sided test

2. Secondary Outcome: Feasibility of Treatment: Number of Participants Completed Treatment According to the Protocol for at Least 24 Weeks
Description: Whether or not the patient completed treatment according to the protocol for at least 24 weeks. Patients who progressed within 24 weeks were considered as not completing.
Time Frame: Baseline to 24 weeks follow-up
Population: Intention to treat population
Measure: Count of Participants; unit: Participants
Arm/Group | A: Nab-Paclitaxel 150 mg/m2 Days 1,15 | B: Nab-Paclitaxel 100 mg/m2 Days 1,8,15 | C: Nab-Paclitaxel 75 mg/m2 Days 1,8,15,22
Number analyzed (Participants) | 83 | 86 | 86
Participants | 40 | 43 | 44

3. Secondary Outcome: Disease Control: Overall Response of Stable Disease for a Duration of ≥24 Weeks
Description: Overall response of stable disease (or non-CR/non-PD for patients with non-measurable disease) for a duration of ≥24 weeks, or better (i.e., partial or complete response) according to RECIST criteria [Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.]
Time Frame: From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 18 months
Population: Intention to treat population
Measure: Count of Participants; unit: Participants
Arm/Group | A: Nab-Paclitaxel 150 mg/m2 Days 1,15 | B: Nab-Paclitaxel 100 mg/m2 Days 1,8,15 | C: Nab-Paclitaxel 75 mg/m2 Days 1,8,15,22
Number analyzed (Participants) | 83 | 86 | 86
Participants | 54 | 59 | 52

4. Secondary Outcome: Best Overall Response
Description: Best response according to RECIST 1.1 criteria [assessed by MRI] recorded from the start of treatment across all time points until end of study treatment. Confirmation of partial or complete response by an additional scan was not requested in this trial.
Time Frame: as for outcome 3
Population: Intention to treat population
Measure: Count of Participants; unit: Participants
Arm/Group | A: Nab-Paclitaxel 150 mg/m2 Days 1,15 | B: Nab-Paclitaxel 100 mg/m2 Days 1,8,15 | C: Nab-Paclitaxel 75 mg/m2 Days 1,8,15,22
Number analyzed (Participants) | 83 | 86 | 86
Participants
  Complete Response (CR) | 5 | 6 | 4
  Partial Response (PR) | 34 | 41 | 35
  Stable Disease (SD)/Non-CR/Non-PD | 39 | 33 | 31
  Progressive Disease (PD) | 3 | 5 | 11
  Not Evaluable (NE) | 2 | 1 | 5

5. Secondary Outcome: Overall Survival
Description: Time from randomization until death from any cause, or censored at date last known alive
Time Frame: Reported after 18.2 months median follow-up since randomization
Population: Intention to treat population
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | A: Nab-Paclitaxel 150 mg/m2 Days 1,15 | B: Nab-Paclitaxel 100 mg/m2 Days 1,8,15 | C: Nab-Paclitaxel 75 mg/m2 Days 1,8,15,22
Number analyzed (Participants) | 83 | 86 | 86
months | 25.8 [16.9 to NA] — Not reported, insufficient number of participants with events. | 26.2 [21.0 to NA] — Not reported, insufficient number of participants with events. | 25.5 [22.7 to NA] — Not reported, insufficient number of participants with events.

6. Secondary Outcome: Changes in Physical Well-being (Change From Day 1 of Cycle 4 to Day 1 of Cycle 6)
Description: Primary quality of life=physical well being; endpoint based on the GLQ 8. The indicator was in Linear Analogue Self-Assessment (LASA) format ranging 0-100 (0=as bad as it can be, 100=as good as it can be).
Time Frame: Assessed from day 1 of cycle 4 through day 1 of cycle 12
Population: Patients who started the maintenance phase of treatment (cycle 4)
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | A: Nab-Paclitaxel 150 mg/m2 Days 1,15 | B: Nab-Paclitaxel 100 mg/m2 Days 1,8,15 | C: Nab-Paclitaxel 75 mg/m2 Days 1,8,15,22
Number analyzed (Participants) | 66 | 72 | 61
units on a scale | -2 [-9 to 5] | 1 [-6 to 7] | 4 [-4 to 11]

ADVERSE EVENTS:
Time Frame: Assessed every 28-day cycle while on treatment and for 30 days after the end of treatment, up to 18 months
Description: Targeted AEs and other grade 3 or higher AEs were collected on CRFs, regardless of attribution.
Arm/Group | A: Nab-Paclitaxel 150 mg/m2 Days 1,15 | B: Nab-Paclitaxel 100 mg/m2 Days 1,8,15 | C: Nab-Paclitaxel 75 mg/m2 Days 1,8,15,22
Serious Adverse Events (participants affected / at risk) | 51/83 | 43/86 | 57/86
Other Adverse Events (participants affected / at risk) | 78/83 | 83/86 | 80/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | A: Nab-Paclitaxel 150 mg/m2 Days 1,15 (N=83) | B: Nab-Paclitaxel 100 mg/m2 Days 1,8,15 (N=86) | C: Nab-Paclitaxel 75 mg/m2 Days 1,8,15,22 (N=86)
Anemia (Blood and lymphatic system disorders) | 5 | 2 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 2 | 2 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 0 | 1
Dry eye (Eye disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 7 | 3 | 2
Ileal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 2 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
Periodontal disease (Gastrointestinal disorders) | 0 | 1 | 0
Stomach pain (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 3
Edema limbs (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 4 | 4 | 9
Fever (General disorders) | 1 | 0 | 0
Multi-organ failure (General disorders) | 1 | 0 | 0
Pain (General disorders) | 3 | 0 | 2
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0 | 0
Bronchial infection (Infections and infestations) | 0 | 0 | 2
Lung infection (Infections and infestations) | 0 | 0 | 1
Nail infection (Infections and infestations) | 0 | 1 | 1
Paronychia (Infections and infestations) | 1 | 0 | 0
Rhinitis infective (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 2 | 1
Skin infection (Infections and infestations) | 0 | 0 | 1
Soft tissue infection (Infections and infestations) | 0 | 1 | 0
Upper respiratory infection (Infections and infestations) | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Wound infection (Infections and infestations) | 0 | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Vascular access complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 18 | 24 | 21
Platelet count decreased (Investigations) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 3 | 0 | 1
Alkaline phosphatase increased (Investigations) | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 3 | 0 | 1
Creatinine increased (Investigations) | 0 | 0 | 1
GGT increased (Investigations) | 3 | 1 | 2
Weight gain (Investigations) | 1 | 0 | 0
White blood cell decreased (Investigations) | 0 | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 3 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal and connective - Other (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Peripheral Sensory Neuropathy (Nervous system disorders) | 7 | 4 | 5
Nervous system disorders - Other (Nervous system disorders) | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 1
Spasticity (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 2 | 0 | 1
Renal and urinary disorders - Other (Renal and urinary disorders) | 0 | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 1
Reproductive system and breast (Reproductive system and breast disorders) | 0 | 1 | 0
Breast pain (Reproductive system and breast disorders) | 1 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 1 | 0
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory thoracic mediastinal - Other,10038738 (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Nail ridging (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Periorbital edema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 5 | 4
Thromboembolic event (Vascular disorders) | 3 | 3 | 4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | A: Nab-Paclitaxel 150 mg/m2 Days 1,15 (N=83) | B: Nab-Paclitaxel 100 mg/m2 Days 1,8,15 (N=86) | C: Nab-Paclitaxel 75 mg/m2 Days 1,8,15,22 (N=86)
Peripheral Sensory Neuropathy (Nervous system disorders) | 51 | 58 | 55
Recurrent Laryngeal nerve Palsy (Nervous system disorders) | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 28 | 35 | 42
Platelet count decreased (Investigations) | 8 | 8 | 4
Anemia (Blood and lymphatic system disorders) | 46 | 55 | 55
Nausea (Gastrointestinal disorders) | 32 | 31 | 40
Vomiting (Gastrointestinal disorders) | 10 | 11 | 17
Diarrhea (Gastrointestinal disorders) | 21 | 28 | 27
Heart Failure (Cardiac disorders) | 0 | 0 | 3
Sinus Tachycardia (Cardiac disorders) | 2 | 4 | 3
Allergic Reaction (Immune system disorders) | 8 | 4 | 4
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-01-06): https://cdn.clinicaltrials.gov/large-docs/25/NCT01746225/Prot_000.pdf
  • Statistical Analysis Plan (2016-03-01): https://cdn.clinicaltrials.gov/large-docs/25/NCT01746225/SAP_001.pdf